CLINICAL TRIAL: NCT05375201
Title: Optimizing Clinical Decision-Making and Virtual Reality Exercise Training in Degenerative Lumbar Spine Disease
Brief Title: Clinical Decision-Making and Virtual Reality Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202003149RINC
Record Dates: First submitted 2022-03-01; First posted 2022-05-16 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-03

CONDITIONS: Degenerative Lumbar Spinal Stenosis; Degenerative Disc Disease; Degenerative Spondylolisthesis; Degenerative Intervertebral Discs
Keywords: virtual reality; degenerative lumbar spine disease; rehabilitation; biomechanic; balance
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- VR skateboarding training (Experimental): specific rehabilitation exercise for improving postural balance
  Interventions: Other: VR skateboarding training

INTERVENTIONS:
Other: VR skateboarding training — The virtual reality skateboard training (VR-skate) is used treadmill-based training. Virtual reality system is integrated into the split-belt treadmill for VR-skate. Participants slide the swing leg (sliding leg) along with the moving treadmill belt at a comfortable speed (same as walking speed).

SUMMARY:
Degenerative lumbar spine disease (DLSD) is common in elderly individuals and can result in pain, muscle weakness, and paresthesia. Numerous studies have reported that patients with DLSD usually have postural balance instability, which may affect the patient's gait, functional activities, and quality of life. The investigators propose to achieve the following aims: (1) to develop a clinical balance diagnostic tool to identify patients with DLSD who may require lumbar surgery (2) to investigate the effects of virtual reality skateboard exercise training on gait and balance in patients with DLSD, as well as to compare them with asymptomatic participants.

ELIGIBILITY:
Inclusion Criteria:

* 1) able to stand and walk for 5 minutes independently
* 2) aged between 50 and 80 years
* 3) received a diagnosis of DLSD based on imaging

Exclusion Criteria:

* 1) previous lumbar surgery
* 2) neurological disorder such as stroke or spinal cord injury
* 3) metabolic disease such as diabetes mellitus
* 4) vestibular disease such as Meniere's disease.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Postural balance | 1 year
  The postural balance measurements are performed by using a force platform. The data from the force platform is used to calculate the mean velocity (unit: cm/s), mean distance (unit: cm), mean frequency (unit: Hz), and 95% confidence ellipse area (unit: cm^2)
Functional assessment | 1 year
  Functional assessment is a process that allows for the identification of disability. The data from the functional assessment is used to calculate walking speed (unit: m/s), walking distance (unit: m), and duration (unit: s).
Muscle activities | 1 year
  Electromyography is a technique for evaluating and recording muscle activity. The data from electromyography is used to calculate a normalized value (unit: ratio).
Kinematic variables | 1 year
  A motion capture system is used to measure the joint kinematics. The data is used to calculate joint angles (unit: degree) and the displacement of the center of mass (unit: cm).
Lumbar Cobb angle | 1 year
  The Lumbar Cobb angle is a measure of the curvature in the lower spine, determined from X-ray images by assessing the angle between the most tilted vertebrae (unit: degree)
Body composition | 1 year
  Body composition was evaluated utilizing the bioelectrical impedance analysis technique. The primary parameters assessed encompassed body fat percentage, visceral fat area, lean muscle mass of the trunk, and the average muscle mass of the lower extremities (unit: percentage %) .
Pain by Visual Analog Scale (VAS) | 1 year
  The VAS pain scale, ranging from 1 to 10, provides a rapid assessment of pain intensity, with individuals marking their level of pain on a line from "no pain" to "worst pain imaginable (unit: score) .
Roland-Morris Disability Questionnaire (RMDQ) | 1 year
  The RMDQ (Roland-Morris Disability Questionnaire) is a widely used self-reported questionnaire that assesses the impact of low back pain on daily functioning. It consists of 24 statements related to daily activities affected by back pain. It's commonly used in clinical settings to evaluate the severity of low back pain and track treatment progress (unit: score). Scores range from 0 to 24, with higher scores indicating more severe disability.

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Li Hsu, Ph.D, Principal Investigator — National Taiwan Unversity
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, 100, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen JH, Chen PJ, Kantha P, Tsai YC, Lai DM, Hsu WL. Examining the influence of body fat distribution on standing balance and functional performance in overweight female patients with degenerative lumbar disease. Front Bioeng Biotechnol. 2024 Jun 21;12:1375627. doi: 10.3389/fbioe.2024.1375627. eCollection 2024. PMID 38974656